CLINICAL TRIAL: NCT04864639
Title: A Transition of Care Model From Hospital to Community for Hispanic/Latino Adult Patients With Diabetes.
Acronym: TOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00103607; 5P30DK111022-05 (NIH)
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Results first posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Spanish; Transition of Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transition of Care (Experimental): Experimental: 32 participants will be discharged to a newly developed discharge/transition of care model.
  Interventions: Other: Transition of Care Model

INTERVENTIONS:
Other: Transition of Care Model — Participants with diabetes, Hispanic/Latinos, adults will receive newly developed discharge instructions.
  Other Names: Patient discharge model

SUMMARY:
This pilot study was designed to address the existing gap in the transition of care of Hispanic/Latino Adults with diabetes from hospital to community. The over arching goal of this study is to develop, test, and determine the feasibility of a transition of care (ToC) model from the hospital to the community for adult Hispanic/Latino patients with diabetes.

DETAILED DESCRIPTION:
This pilot study is designed to develop, test, and determine the feasibility of a transition of care model from the hospital to the community for adult Hispanic/Latino patients with diabetes. The proposed study originally designed was randomized pilot study with two arms: 1) the usual transition of care and (2) a transition of care model newly developed using information collected during our study aim 1. Given the multiple challenges brought on by the COVID-19 pandemic, we found it necessary to adapt and modify the original study design. The study designed with approval from our funding team was changed to utilize the Plan-Do-Act-Study (PDSA) as a framework. The PDSA is an iterative process that allows us to test on a small scale and document unexpected observations and determine what modifications should be made and prepare for next test. A transition of care (ToC) model will be developed based on the following data: 1) results from semi-structure interviews from our first cohort of Hispanic/Latino participants with diabetes recently discharged from the hospital and providers from the hospital and community ; 2) feedback from participants in the community during the Community Consultation Studio . Once developed, the ToC model will be tested with a total of 16 participants discharged from the hospital to the community. The model will incorporate the preference and perspective of providers and patients. Participants will complete a set of of questionnaires (demographic, sociocultural and medical history) prior to discharge and a follow up telephone call interview 30-days post discharge. A total of 5 participants for the first set of participants will be interview. These interviews will be analyzed for common patterns and themes for which the results will inform improvement of the ToC. A second cohort of participants (n=16) will be enrolled. And complete the same set of questionnaires along with the 30 day post discharge telephone call. Finally, after implementing and enrolling the second cohort, as small subset will be interview including providers (n=3) to obtain additional information that will inform further improvement of the ToC.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosis of Diabetes Mellitus
* Self-identified Hispanic/Latino
* Spanish or English speaking
* Currently hospitalized in the Duke University Health System
* Able to provide informed consent without a proxy

Exclusion Criteria:

* There is no exclusion criteria based on comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonor Corsino, MD, Principal Investigator — Duke University
Locations (1):
- Leonor Corsino, MD, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that results reported in manuscript after deidentification (text, tables, figures, appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Sharing will end 5 years after manuscript publication

REFERENCES:
- [Derived] Corsino L, Padilla BI. A transition of care model from hospital to community for Hispanic/Latino adult patients with diabetes: design and rationale for a pilot study. Pilot Feasibility Stud. 2022 Dec 5;8(1):246. doi: 10.1186/s40814-022-01203-z. PMID 36471392

RESULTS

PARTICIPANT FLOW:
Groups:
- Transition of Care: Experimental: Participants will be discharged to a newly developed discharge/transition of care model.
  Transition of Care Model: Participants with diabetes, self-identified Hispanic/Latinos, adults will receive newly developed discharge instructions.
Period: Overall Study
Arm/Group | Transition of Care
Started | 12
Completed | 10
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transition of Care
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Emergency Department (ED) Visits Within 30 Days Post Discharge
Description: The number of times the participant has revisited the ED after their discharge from the hospital.
Time Frame: 30 days post-discharge
Measure: Mean (Standard Deviation); unit: emergency department visits
Arm/Group | Transition of Care
Number analyzed (Participants) | 12
emergency department visits | 0 (0)

2. Secondary Outcome: Unplanned Readmissions to the Hospital Within 30 Days Post Discharge
Description: The number of times the patient is readmitted to the hospital for unplanned admissions after discharge.
Time Frame: up to 30 days
Measure: Mean (Standard Deviation); unit: hospital readmissions
Groups:
- Transition of Care: Experimental: Participants will be discharged to a newly developed discharge/transition of care model.
  Transition of Care Model: Participants with diabetes, Hispanic/Latinos, adults will receive newly developed discharge instructions.
Arm/Group | Transition of Care
Number analyzed (Participants) | 12
hospital readmissions | 0 (0)

ADVERSE EVENTS:
Time Frame: Approximately 30 days
Arm/Group | Transition of Care
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Given the multiple challenges brought on by the COVID-19 pandemic, the PIs found it necessary to modify the original study design. Under the guidance of the study sponsors/mentors, the study design was changed to a Plan-Do-Study-Act (PDSA) cycle framework. The rationale for this modified approach was informed by the fact that "the usual transition of care" was significantly altered during the pandemic. The recruitment goal was not reached before running out of funding for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT04864639/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT04864639/ICF_000.pdf